CLINICAL TRIAL: NCT06588010
Title: Multicentre Randomised Double-blind Superiority Trial With a Roll-over Phase to Assess the Efficacy of OM-89 vs Placebo in Reducing Antibiotic Consumption Associated With the Treatment of Urinary Tract Infections in Patients With Neurogenic Bladder
Brief Title: Assess the Efficacy of OM-89 vs Placebo in Reducing Antibiotic Consumption Associated With the Treatment of Urinary Tract Infections in Patients With Neurogenic Bladder
Acronym: RETRAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PIROTH OMPharma 2023
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — OM 89

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients in the experimental arm (Experimental)
  Interventions: Drug: OM-89 [Uro-Vaxom® Capsule] OM-89 placebo [Uro-Vaxom® Capsule placebo]
- Patients in the control arm (Active Comparator)
  Interventions: Drug: OM-89 [Uro-Vaxom® Capsule]

INTERVENTIONS:
Drug: OM-89 [Uro-Vaxom® Capsule] — 1st phase and 2nd phase : 1 capsule per day of OM-89 for 90 consecutive days followed by a period of 90 days without treatment, then one capsule per day of OM-89 for 10 consecutive days each month for three months.
  Arms: Patients in the control arm
Drug: OM-89 [Uro-Vaxom® Capsule] OM-89 placebo [Uro-Vaxom® Capsule placebo] — 1st phase: 1 capsule per day of placebo for 90 consecutive days followed by a period of 90 days without treatment, then one capsule per day of placebo for 10 consecutive days each month for three months.
  Then 2nd phase: 1 capsule a day of OM-89, for 90 consecutive days followed by a period of 90 days without treatment, then one capsule a day of OM-89 6mg for 10 consecutive days each month for three months.
  Arms: Patients in the experimental arm

SUMMARY:
Recurrent urinary tract infections (UTIs) in patients with a neurogenic bladder using clean intermittent catheterization (CIC) are a major problem. In this population, urinary tract infections are the most frequent cause of morbidity and the second leading cause of mortality (Buzzell A, Spinal Cord, 2020). It is also the leading cause of healthcare use and consumption (A. Dinh, MMI 2019). In addition, multidrug-resistant bacteria (MRB) are frequently implicated, accounting for up to 50% of cases (Samal V BMC Infect Dis 2022, A. Dinh Spnal cord 2016), due to high exposure to antibiotics and frequent and prolonged hospitalisations.

The very frequent recurrence of urinary tract infections encourages exposure to antibiotics, so prevention is of vital importance. Prevention based on treatments other than antibiotics (non-antibiotic prophylaxis) is of the greatest interest, not only to prevent UTIs, but also to reduce exposure to antibiotics and the ecological pressure they exert. However, few strategies are available, and very few have been well evaluated in high-risk populations.

Bacterial lysates such as Escherichia Coli extract (OM-89), an immunoactive prophylaxis, are an original and innovative strategy that has been developed for the prevention of recurrent UTIs, and could constitute a therapeutic option in particularly at-risk populations.

In vivo studies have shown that OM-89 :

* increases IgA levels in intestinal secretions and in the urine of mice (Bosh AV Immunopharmacol Immunotoxicol 1988; Baier W Arzneim Forsch Drug Res 1997),
* stimulates the production of serum IgG and IgA recognising a number of bacteria isolated from patients with urinary tract infections and enterohaemorrhagic E. coli infections (Huber M, Int J immunopharmacol 2000),
* stimulates the killing capacity of rabbit polymorphonuclear leukocytes against E. coli and S. aureus (Nauck M, Int J Exp Clin Chemother 1991),
* protects against acute infection with E. coli or P. aeruginosa,
* and inhibits inflammation associated with lipopolysaccharide-induced cystitis in mice (Lee SJ, World J Urol 2006).

Clinically, certain studies in patients with recurrent UTIs have shown a significant reduction in the number of urinary tract infections with OM-89 compared to placebo or an antibiotic (Bauer Eur Urol 2005; Naber KG Int J Antimicrob Agents 2009; Wade DT, Clin Rehabil 2020).

However, these promising results suffer from methodological limitations and need to be confirmed by a high-quality trial carried out on a sample appropriate to the research question and in a homogeneous patient population.

Patients with spinal cord injuries are a population at high risk of recurrent UTIs, and prevention is a major issue, given the incidence of MRBs in this population. It is therefore important in this high-risk population not only to rigorously evaluate the efficacy of OM-89 in reducing antibiotic consumption for UTIs, but also to assess its impact on bacterial resistance and on the microbiota (urinary and digestive). These patients could therefore see significant benefits: less frequent urinary tract infections and reduced antibiotic use. In addition, this population could serve as a model for other populations with or without neurological impairment suffering from recurrent UTIs

ELIGIBILITY:
Inclusion Criteria:

* Person who has given written consent
* Patient aged 18 years or older
* Patient with a stabilised neurogenic bladder following spinal cord injury thaht has not progressed for more than 2 years and who has undergone a urodynamic examination in the last 2 years.
* Patients using CIC (5 to 6 per day)
* Patients who have received at least 6 courses of antibiotic treatment for UTIs in the 12 months prior to screening (whether for curative or prophylactic reasons)
* Patients with a negative urine culture between screening visit and randomisation or treated with antibiotics for urinary decontamination prior to randomisation.

Exclusion Criteria:

* Person who is not affiliated with the national health insurance system
* Person subject to a measure of legal protection (guardianship, tutorship)
* Person subject to a court order
* Adults unable to express consent
* Patients using a urinary drainage method other than CIC
* Patients with urinary lithiasis at the time of inclusion (assessed by renal imaging in the previous year as part of routine management for patients with a history(s) of lithiasis or within 3 years for patients with no history)
* Presence of an endo-urinary device (urinary prosthesis, ureteral stent)
* Enterocystoplasty or irradiated bladder (past or present)
* Known allergy or previous intolerance to the active substance or one of the excipients of OM-89 or placebo
* Patient requiring ongoing or short-term prolonged antibiotic therapy (e.g. infected bedsore, etc.)
* Patient treated with bacterial lysates (including OM-89) in the 6 months prior to randomisation
* Unable or unwilling to stop prophylactic antibiotic therapy prior to randomisation
* Patient with a known malignant tumour or neoplasia
* Patient with an autoimmune disease
* Patient treated with long-term or bolus corticosteroids, anti-CD20 and anti-rejection therapy in the 6 months prior to screening
* Patient currently taking part in another study on an investigational device or drug related to urinary tract infections, or who has received another investigational treatment in the 30 days prior to screening.
* Patient unable to collect information in a daily diary.
* Patient unable to understand follow-up by telephone.
* Patients planning to move to another residence in the year following randomisation
* Non-menopausal women who are not surgically sterile (bilateral oophorectomy or hysterectomy) AND pregnant, breast-feeding who are declare that they are planning to conceive at inclusion, or not using effective* contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of antibiotic treatment episodes for UTIs per person-days at risk during the first year. | 12 months
  An episode of treatment is defined as a single prescription of a given antibiotic, regardless of its intended duration (curative or prophylactic). A day at risk is defined as a follow-up day without antibiotic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France